CLINICAL TRIAL: NCT00000602
Title: Pediatric Hydroxyurea in Sickle Cell Anemia (PED HUG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 315; P60HL015157 (NIH); P60HL028391 (NIH); P60HL020985 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2005-10

CONDITIONS: Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies | interventions — Hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea

SUMMARY:
To determine whether hydroxyurea prevents the onset of chronic end organ damage in young children with sickle cell anemia.

DETAILED DESCRIPTION:
BACKGROUND:

Sickle cell anemia is a complex syndrome with multiple organ system disturbances brought about by the interplay of genetic, humoral, vascular and environmental factors. The clinical course can be one of abrupt and insidious exacerbations and remissions, often migratory and repetitive. These events may result in impairment of function, permanently damaged organs, and ultimately death. Although there is wide variability in the clinical expression of sickle cell disease, this complex set of clinical manifestations is experienced by most patients. In addition, there is no evidence that the primary disease process is different in children when compared with adults with regard to painful episodes. However, children have a higher incidence of respiratory viral infections, and are susceptible to pneumococcal septicemia. With the successful completion of the Multicenter Study of Hydroxyurea (MSH) Trial in adults, attention has now been focused on the use of this agent in children.

The Cooperative Study of Sickle Cell Disease (CSSCD) has demonstrated that sickle cell anemia patients with increased painful episode rates die at a younger age. In addition, increased levels of fetal hemoglobin are associated with improved survival, and is probably a reliable childhood forecaster of adult life expectancy. The beneficial effect produced by hydroxyurea is thought to occur because it increases fetal hemoglobin levels. Therefore, if chronic end organ damage can be prevented in early childhood by hydroxyurea administration, and if the crisis rate can be decreased by hydroxyurea use early in life, sickle cell anemia patients may experience increased longevity and an improved quality of life.

DESIGN NARRATIVE:

The Phase I-Phase II study, HUG-KIDS, examined the safety of hydroxyurea. Children with sickle cell anemia, age 5 to 15 years, were eligible for this multicenter Phase I/II trial. Hydroxyurea was started at 15 mg/kg/d and escalated to 30 mg/kg/d unless the patient experienced laboratory toxicity. Patients were monitored by 2-week visits to assess compliance, toxicity, clinical adverse events, growth parameters, and laboratory efficacy associated with hydroxyurea treatment. Eighty-four children were enrolled between December 1994 and March 1996. Sixty-eight children reached maximum tolerated dose (MTD) and 52 were treated at MTD for 1 year. The study was conducted at four Comprehensive Sickle Cell Centers by the following investigators: Thomas R. Kinney at Duke University Medical Center, Durham, North Carolina; Kwaku Ohene-Frempong at Children's Hospital of Philadelphia; Orah S. Platt at Children's Hospital in Boston; and Elliot Vichinsky at Children's Hospital in Oakland, California. The complete study lasted three years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Children with sickle cell disease and between the ages of five and eighteen years.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1994-04; Study Completion 1997-03 (Actual)

REFERENCES:
- [Background] Phase I/II Multicenter Pediatric Trial of Hydroxyurea (HUG-Kids). Blood, 90 (Suppl 1):Abstract # 1974, 1997.
- [Background] Kinney TR, Helms RW, O'Branski EE, Ohene-Frempong K, Wang W, Daeschner C, Vichinsky E, Redding-Lallinger R, Gee B, Platt OS, Ware RE. Safety of hydroxyurea in children with sickle cell anemia: results of the HUG-KIDS study, a phase I/II trial. Pediatric Hydroxyurea Group. Blood. 1999 Sep 1;94(5):1550-4. PMID 10477679
- [Background] Wang WC, Helms RW, Lynn HS, Redding-Lallinger R, Gee BE, Ohene-Frempong K, Smith-Whitley K, Waclawiw MA, Vichinsky EP, Styles LA, Ware RE, Kinney TR. Effect of hydroxyurea on growth in children with sickle cell anemia: results of the HUG-KIDS Study. J Pediatr. 2002 Feb;140(2):225-9. doi: 10.1067/mpd.2002.121383. PMID 11865275